CLINICAL TRIAL: NCT03798821
Title: Nutritional Clinical Trial to Evaluate the Antioxidant Efficacy of a Product Probiotic in Research
Brief Title: The Antioxidant Efficacy of a Product Probiotic in Research
Acronym: BIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCAM-CFE-0003
Record Dates: First submitted 2018-03-15; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — maltodextrin; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): One capsule a day will be consumed. At breakfast for the six weeks.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus, Lactobacillus casei y Bifidobacterium longum (100MG); Dietary Supplement: Lactobacillus rhamnosus, Lactobacillus casei y Bifidobacterium longum (300MG)
- Comparator (Placebo Comparator): One capsule a day will be consumed. At breakfast for the six weeks.
  Interventions: Dietary Supplement: maltodextrin and sucrose (PLACEBO)

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus, Lactobacillus casei y Bifidobacterium longum (100MG) — six weeks of consumption
  Arms: Experimental
Dietary Supplement: Lactobacillus rhamnosus, Lactobacillus casei y Bifidobacterium longum (300MG) — six weeks of consumption
  Arms: Experimental
Dietary Supplement: maltodextrin and sucrose (PLACEBO) — six weeks of consumption
  Arms: Comparator

SUMMARY:
Determine the efficacy of the investigational product versus placebo in reducing stress oxidative during the performance of a physical exercise of a certain intensity and duration.

DETAILED DESCRIPTION:
The effectiveness of a probiotic for oxidative stress after eight weeks of the product to study will be checked. the sample will be formed by cyclists that will submit to a baseline exercise and after the product is taken.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 45 years
* Sex: male, of Caucasian race, selected from the general population.
* Subjects that perform aerobic physical exercise between 2 and 4 times a week.
* Volunteers capable of understanding the clinical study, willing to grant consent informed in writing and to comply with the procedures and requirements of the study

Exclusion Criteria:

* Subjects with a history of any chronic disease.
* History of bronchial asthma or chronic obstructive pulmonary disease, disease Reactive airways such as bronchial asthma, a history of bronchial asthma or severe chronic obstructive pulmonary disease.
* Sinus bradycardia, second or third degree of atrioventricular block, insufficiency manifest cardiac or cardiogenic shock.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Participation in another clinical trial in the three months prior to the study Lack of will or inability to comply with clinical trial procedures.
* Subjects diagnosed and / or under treatment for arterial hypertension.
* Smoking subjects (> 10 cigarettes a day).
* Subjects with body mass index greater than 35 Kg / m2 (BMI> 30).
* Subjects with a history of drug, alcohol or other substance abuse or other factors that limit their ability to cooperate during the study.
* Subjects whose condition does not make them eligible for the study according to the researcher's criteria.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Oxidative damage to lipids | Oxidative lipid damage will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  It will be measured by isoprostanes in urine 24 hours.

SECONDARY OUTCOMES:
Oxidative damage to DNA | Oxidative damage to DNA will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  Analysis of 8-oxo 2'-deoxyguanosine in 24-hour urine.
Oxidative damage to proteins. | Oxidative damage to protein will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  Analysis of serum carbonyl groups
Oxidative damage to lipids | Oxidative damage to lipids will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  analysis of malondialdehyde in plasma
Blood analysis | Blood analysis will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  serum carbonyls. It is measured in nmol / mg proteins
Blood analysis | Blood analysis will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  Malondialdehyde in plasma
Blood analysis | Blood analysis will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  Oxidized LDL.
Blood analysis | Blood analysis will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  Antioxidant capacity.
Blood analysis | Blood analysis will be measured by the ELISA test on two different occasions. The measurements will be made at the beginning and at six weeks of consumption of the product.
  glutathione metabolism. It is measured in nmol / mg proteins

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez Macarro M, Avila-Gandia V, Perez-Pinero S, Canovas F, Garcia-Munoz AM, Abellan-Ruiz MS, Victoria-Montesinos D, Luque-Rubia AJ, Climent E, Genoves S, Ramon D, Chenoll E, Lopez-Roman FJ. Antioxidant Effect of a Probiotic Product on a Model of Oxidative Stress Induced by High-Intensity and Duration Physical Exercise. Antioxidants (Basel). 2021 Feb 22;10(2):323. doi: 10.3390/antiox10020323. PMID 33671691